CLINICAL TRIAL: NCT01532180
Title: A Pilot Study and Follow Up of the Use of a Hypoglossal Nerve Implant for Treatment of Obstructive Sleep Apnea
Brief Title: Safety and Efficacy of a Hypoglossal Nerve Implant for the Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ImThera Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: LivaNova (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMT 2009-01/02/03
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Respiration Disorders; Signs and Symptoms, Respiratory; Syndrome, Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea, neurostimulation, hypoglossal nerve
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Respiration Disorders; Signs and Symptoms, Respiratory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- THN Therapy (Experimental)
  Interventions: Device: aura6000 System

INTERVENTIONS:
Device: aura6000 System — The aura6000 device is an implanted hypoglossal nerve stimulator designed to maintain wakeful muscle tone of the tongue during sleep. It is implanted through a short surgical procedure. The implant is programmed to provide the optimal stimulation parameters for the patient. The therapy is controlled by a hand-held remote control allowing the patient to start, stop, and pause the therapy during times of sleep.

SUMMARY:
The objective of the study is to determine the safety and preliminary efficacy in patients utilizing the aura6000 System for the treatment of Obstructive Sleep Apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe obstructive sleep apnea (AHI 15 to 60).
* Cannot or will not tolerate CPAP treatment.
* Body mass index (BMI) between 25 and 40
* Able to read, understand, sign and date the written informed consent form

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mean change in AHI measured through in-lab polysomnography (PSG) compared to baseline. | 3 and 12 months post-implant
Adverse events and Serious Adverse events peri and post-operatively | 3 and 12 months post-operative

SECONDARY OUTCOMES:
Mean change in Quality of Life outcomes measured with ESS (Epworth Sleepiness Scale) as compared to baseline. | 3 and 12 months post-operative
Mean change in Quality of Life outcomes measured with FSS (Fatigue Severity Scale) as compared to baseline. | 3 and 12 months post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rodenstein, MD, Principal Investigator — Clinique Univ. Saint-Luc
Locations (1):
- Clinique Univ. Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Mwenge GB, Rombaux P, Dury M, Lengele B, Rodenstein D. Targeted hypoglossal neurostimulation for obstructive sleep apnoea: a 1-year pilot study. Eur Respir J. 2013 Feb;41(2):360-7. doi: 10.1183/09031936.00042412. Epub 2012 May 17. PMID 22599356